CLINICAL TRIAL: NCT04205513
Title: Randomized Controlled Trial of a Mobile Phone-based Telemonitoring Application Utilized for the Facilitation of Medication Titration for Patients With Heart Failure
Brief Title: Use of Telemonitoring to Facilitate Heart Failure Medication Titration
Acronym: Medly Titrate
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-5351.0; RGPIN-2014-04486 (Other Grant/Funding Number: Natural Sciences and Engineering Research Council of Canada)
Record Dates: First submitted 2018-11-21; First posted 2019-12-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure
Keywords: Telemonitoring; Titration; Remote monitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Standard titration management strategy, consisting of regular in-office visits.
- Study Group (Experimental): Remote titration management strategy, consisting of telephone contacts, which will utilize data from the Medly system.
  Interventions: Device: Medly

INTERVENTIONS:
Device: Medly — Medly is a mobile phone-based telemonitoring system that enables patients with heart failure to take clinically relevant physiological measurements with wireless home medical devices and answer symptom questions on the mobile phone. The measurements are automatically and wirelessly transmitted to the mobile phone and then to a data server.
  Arms: Study Group

SUMMARY:
Heart failure (HF) is a common diagnosis with high prevalence, reduced life expectancy and a significant clinical and economic burden. Large-scale randomized controlled trials have demonstrated that combination drug therapy, optimized to maximal tolerated doses, improves clinical outcomes in HF patients. However, evidence suggests that in clinical practice many patients never achieve target doses.

Barriers to medication titration include provider and patient-related factors, as well as limited time and support facilities to enable regular monitoring. Telemonitoring is a potential component in the management of HF that can provide reliable and real-time physiological data for clinical decision support, alerting, and patient self-management.

The primary objective of this study is to evaluate the effectiveness and safety of the implementation of telemonitoring to facilitate HF medication titration. The secondary objective is to obtain a deeper understanding of the experience of clinicians and HF patients taking part in the remote titration program.

The study will be conducted at the Peter Munk Cardiac Centre (PMCC), University Health Network, in Toronto. It will be based on a mixed methods effectiveness-implementation hybrid design and incorporate process evaluations alongside assessment of clinical outcomes.

The effectiveness research component will be assessed via a 2-arm randomized controlled trial (RCT), which will enroll 108 patients in total. The RCT will compare a predefined remote titration management strategy, which will utilize data from a smartphone-based telemonitoring system, with a standard titration management strategy consisting of regular in-office visits, and assess the efficacy and safety of the telemonitoring system in facilitating titration.

The implementation research component will consist of a qualitative study based on semi-structured interviews with a purposive sample of clinicians and patients, and assess the factors that can positively impact the implementation and effectiveness of the intervention.

DETAILED DESCRIPTION:
BACKGROUND Heart failure (HF) is a common diagnosis affecting at least 26 million people worldwide. Based on available data from the US and Europe, the overall prevalence of HF ranges from 1% to 12%. The lifetime risks of developing HF, assessed and reported based on a large, diverse, multi-cohort group of 39,578 participants, was shown to be about 30% to 42% in white men, 20% to 29% in black men, 32% to 39% in white women, and 24% to 46% in black women. Survival rates reported in studies also varied, with data from the US and Europe indicating a 1-year survival rate of 89% to 70%, and 5-year survival rates ranging from 59% to as low as 35%, reflecting a significant increase in the risk of death compared to the general age and gender matched population.

The discrepancies in the estimates can most likely be attributed to differences in patient selection, as well as ascertainment and adjustment approaches, however, irrespective of the precise rates, several trends are congruent across studies, including high prevalence, reduced life expectancy, worsening profile with aging and, at best, stagnant incidence rates over the last several decades. These trends have tremendous implications since HF patients are major consumers of healthcare resources.

Large-scale randomized controlled trials have demonstrated that angiotensin receptor-neprilysin inhibitors, angiotensin-converting enzyme inhibitors (ACEIs), angiotensin receptor blockers (ARBs), beta-blockers and mineralocorticoid receptor antagonists all improve clinical outcomes in HF patients, suggesting that their combination could translate to a 60-70% relative risk reduction in all-cause mortality, and clinical guidelines recommend up titrating the treatments to maximal tolerated doses. However, in clinical practice, evidence from 12,440 HF patients of the European Society of Cardiology Heart Failure Long-Term Registry, showed that about 30% of patients were on target doses of ACEIs, 18% were on target doses of beta-blockers, and approximately one-third had no documented reason for the failure to up-titrate. Barriers to medication titration include health-provider knowledge, self-efficacy and attitudes, patient-related factors and limited time and support facilities to enable regular monitoring.

Remote patient monitoring is a potential component in the management of HF that can provide reliable and real-time physiological data for clinical decision support, alerting, and patient self-management. Telemonitoring enables patients to track their vital signs and symptoms, and also to receive automated instruction and clinical intervention during "teachable moments" (i.e., clear actions are provided when the context is most appropriate). The automated instructions are based on current physiological measurements, self-monitored symptoms, and can be readily analyzed. Automated real-time alerts and frequently collected and analyzed physiological/symptom data can also support clinical decisions by healthcare providers. Several previous studies, including 2 studies conducted by the same research team, have shown that the use of telemonitoring interventions for the management of chronic conditions can lead to positive health outcomes and significant reductions in healthcare costs if the intervention is designed and implemented appropriately. Telemonitoring for HF patients has been shown to be particularly beneficial, demonstrating reduced mortality (risk ratio=0.64; 95% confidence interval: 0.48-0.85), reduction in the use of health services, and similar or improved quality of life and satisfaction compared with standard care.

In response to this evidence, Medly, a telemonitoring program for patients with Heart Failure (HF) has been launched at the University Health Network (UHN). This program is integrated into the Ted Rogers Centre of Excellence in Heart Function at the Peter Munk Cardiac Centre (PMCC) as part of the standard of care.

OBJECTIVES The primary objective of this study is to evaluate the effectiveness and safety of the implementation of telemonitoring to facilitate HF medication titration and its impact on.

The telemonitoring titration management strategy will be compared to the standard titration management program consisting of regular in-office visits.

The hypothesis underlying the primary objective of the study is that both management strategies will enable a comparable proportion of patients to reach optimal doses of HF medications, within similar timeframes, but that telemonitoring will significantly reduce the cost of healthcare resource utilization and patient burden.

The secondary objective of this study is to obtain a deeper understanding of the experience of clinicians and HF patients taking part in the remote titration program, in order to develop better awareness of the factors that can positively impact the implementation and effectiveness of the intervention.

The mobile phone-based telemonitoring system (Medly) enables patients with HF to take clinically relevant physiological measurements with wireless home medical devices in addition to answering symptom questions on the mobile phone. The measurements are automatically and wirelessly transmitted to the mobile phone and then to a data server. Specifically, patients monitor daily weight, blood pressure/heart rate, symptoms, and some patients monitor their activity as determined by their cardiologist. Automated self-care instructions/messages that have been carefully developed with healthcare specialists are sent to the patient based on the readings and reported symptoms. If there are signs of their status deteriorating, an alert is sent to a clinician at the Heart Function Clinic. Through a secure web portal, clinicians receive all relevant patient data, thereby granting them access to current trends and historic data reported by their patients. Clinicians will use information provided by Medly to facilitate remote titration of HF medication doses. A predefined titration management strategy will be established during the initial clinic visit, in accordance with HF management guidelines. Subsequently, telephone contacts will take place at 2-week intervals to titrate medication doses, based on patient-reported data.

PATIENT DATA ACQUISITION Patients will be followed for the duration of their time in the Medly Titrate Program. Data acquisition will include telemonitoring data, patient lab test and examination results, application usage data, data regarding healthcare utilization.

All patients randomized into the study group will also be invited to participate in individual interviews intended to assess their experiences and perceptions regarding the Program upon titration completion.

PROVIDER AND PROGRAM STAFF DATA ACQUISITION Healthcare providers and program staff will be asked to participate in interviews to determine their perceptions of the Medly Titrate Program and of its implementation within existing clinic services.

DATA ANALYSIS Descriptive statistics will be run regularly on all patient outcome measures to monitor the program for quality improvement purposes. Parametric and non-parametric tests will be performed to compare data at baseline and titration completion.

Statistical analyses will be performed using the statistical software application SPSS. Interview data will be analyzed using a conventional content analysis approach. Two evaluators will analyze the transcripts independently and discuss their findings until a consensus is reached. The software program NVivo will be used to help organize the transcript data for analysis.

The underlying assumption is that both remote titration and standard in-office visits will yield similar clinical outcomes, but that the remote management strategy will significantly reduce healthcare resource utilization. Therefore, non-inferiority and superiority analyses will be performed. The intention-to-treat-population, which will include all randomized patients, shall be the study population used for the non-inferiority analysis. The per-protocol-population, which will include all patients who have been treated according to protocol, excluding those who: (a) demonstrated inadequate compliance, or (b) withdrew randomized therapy prematurely without cause, shall be the study population used for the superiority analysis.

DISSEMINATION STRATEGY Results will be shared with Medly Program and HF Clinic decision-makers as they become available, as they will be used for quality improvement purposes. In addition, as these results will be of interest to other clinical settings intending to implement similar telemonitoring programs, the investigators plan to disseminate findings through publications in appropriate scientific journals and through presentations at scientific conferences, as well as other relevant media avenues (e.g., news reports).

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to provide informed consent to participate in the program.
* Adult patients (age 18 years or older)
* Diagnosed with HF and followed by a cardiologist at the PMCC Heart Function Clinic, who has primary responsibility for management of the patient's HF.
* New York Heart Association (NYHA) Class II-III.
* Left ventricular ejection fraction (LVEF) 40% or less, based on echocardiography, determined within 3 months prior to randomization.
* Stable HF defined as no hospitalization within 3 months.
* Patient is not yet at target doses of guideline directed medical therapy (ACE inhibitor, and/or angiotensin receptor blocker, and/or b-blocker, and/or mineralocorticoid receptor antagonist at sub-optimal doses), and hence qualifies for up-titration. At the physician's estimate, the patient will require a minimum of about 2 months to achieve target doses of all HF medications
* Patient or their informal caregiver speaks and reads English adequately to participate in the program and understand the alerts/prompts in the Medly application.
* Ability to comply with using Medly (e.g., able to stand on the weight scale, able to answer symptom questions, etc.).

Physicians at the clinics will ultimately determine which patients they believe may benefit from participating in the Medly Titrate Program. For these patients, the Titrate program will be offered in addition to their usual care at the UHN, which includes Medly telemonitoring.

Exclusion Criteria:

Patients will be excluded from the study based on the clinical judgment of their healthcare provider. In addition, the following criteria will exclude patients from participation in the Medly Titrate Program:

* Active acutely decompensated heart failure.
* Already on target doses of guideline-directed medical therapy (GDMT).
* Inability to titrate medications due to adverse events including:

  * History of angioedema
  * Uncontrolled hypertension
  * Hypotension preventing up-titration
  * Heart rate at rest <56 beats per minute
* Congenital heart disease.
* Previous heart transplant or currently awaiting heart transplant.
* Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid, or other major cardiovascular surgery, PCI, or carotid angioplasty within 6 weeks prior to randomization.
* Obstructive or restrictive cardiomyopathy.
* Second or third degree atrioventricular block without a pacemaker.
* Presence of hemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation.
* Presence of other hemodynamically significant obstructive lesions of the LV outflow tract, including aortic and subaortic stenosis.
* Evidence of hepatic impairment defined as ALAT or ASAT value >three-fold the upper normal limit. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 at randomization or >35% decline in eGFR between visits.
* Known stenosis of both renal arteries.
* Hyper- or hypothyroidism not controlled by treatment.
* Hyperkalemia >5.5 mmol/L at randomization.
* Hyponatremia <130 mmol/L at randomization.
* History of severe asthma or pulmonary disease.
* Presence of any other disease, which in the clinician's opinion would exclude the patient from the study or with a life expectancy of <1 year.

Compliance will be closely monitored to ensure the safety of the patients. As telemonitoring will partially replace clinic visits, adherence to program requirements in terms of physiological measurements and symptom reporting will be necessary to ensure prompt identification of potential side effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving GDMT titration completion | 6 months from enrolment
  The proportion of patients achieving GDMT titration completion at 6 months. (Revised primary outcome, after internal pilot, therefore, 0.025 significance value to be used.)
The number of clinic visits required to achieve GDMT titration completion | Through study completion, an average of 1 year
  The number of clinic visits (either in-person or virtually) required to achieve GDMT titration completion

SECONDARY OUTCOMES:
Median time to GDMT titration completion | Through study completion, an average of 1 year
  Median time to dose optimization
Patient health outcomes (LVEF) | Through study completion, an average of 1 year
  LVEF - Left ventricular ejection fraction, assessed via medical imaging
Patient health outcomes (BNP - Brain natriuretic peptide) levels | Through study completion, an average of 1 year
  BNP (brain natriuretic peptide) levels, assessed via a blood test
Patient health outcomes (Clinical) | Through study completion, an average of 1 year
  Need for hospitalization; HF hospitalization; urgent clinic or emergency department visit
Implementation barriers | Through study completion, an average of 1 year
  Barriers to implementation identified via qualitative research methods (thematic analysis of interviews)
Implementation facilitators | Through study completion, an average of 1 year
  Facilitators of implementation identified via qualitative research methods (thematic analysis of interviews)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Seto, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Artanian V, Rac VE, Ross HJ, Seto E. Impact of Remote Titration Combined With Telemonitoring on the Optimization of Guideline-Directed Medical Therapy for Patients With Heart Failure: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Oct 13;9(10):e19705. doi: 10.2196/19705. PMID 33048057
- [Background] Artanian V, Ross HJ, Rac VE, O'Sullivan M, Brahmbhatt DH, Seto E. Impact of Remote Titration Combined With Telemonitoring on the Optimization of Guideline-Directed Medical Therapy for Patients With Heart Failure: Internal Pilot of a Randomized Controlled Trial. JMIR Cardio. 2020 Nov 3;4(1):e21962. doi: 10.2196/21962. PMID 33141094
- [Derived] Elfassy MD, Runeckles K, Simms N, Anderson GM, Simard A, Brahmbhatt DH, Seto E, Lipscombe A, Faroutan F, Miller FA, Ross HJ; Medly Titrate Study Team. Carbon and Travel Cost Reduction From Remote Medication Titration for Advanced Heart Failure: A Secondary Analysis of a Randomized Controlled Trial. Can J Cardiol. 2025 Dec;41(12):2451-2459. doi: 10.1016/j.cjca.2025.07.026. Epub 2025 Jul 29. PMID 40744126
- [Derived] Brahmbhatt DH, Ross HJ, O'Sullivan M, Artanian V, Mueller B, Runeckles K, Steve Fan CP, Rac VE, Seto E; Medly Titrate Study Team. The Effect of Using a Remote Patient Management Platform in Optimizing Guideline-Directed Medical Therapy in Heart Failure Patients: A Randomized Controlled Trial. JACC Heart Fail. 2024 Apr;12(4):678-690. doi: 10.1016/j.jchf.2024.02.008. PMID 38569821
- [Derived] Artanian V, Ware P, Rac VE, Ross HJ, Seto E. Experiences and Perceptions of Patients and Providers Participating in Remote Titration of Heart Failure Medication Facilitated by Telemonitoring: Qualitative Study. JMIR Cardio. 2021 Nov 25;5(2):e28259. doi: 10.2196/28259. PMID 34842546